CLINICAL TRIAL: NCT00123578
Title: GHB: Effects, Withdrawal and Treatment
Brief Title: GHB Withdrawal Symptoms and Effectiveness of Treatment With Lorazepam Versus Pentobarbital - 1
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Unable to recruit adaquate number of GHB dependent subjects
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Karen Miotto, Clinical Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIDA-14291-1; K23DA014291 (NIH)
Record Dates: First submitted 2005-07-22; First posted 2005-07-25 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Lorazepam; Pentobarbital

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lorazepam (Experimental): Lorazepam for the treatment of mild GHB withdrawal.
  Interventions: Drug: Lorazepam
- Pentobarbital (Active Comparator): Pentobarbital for the treatment of mild GHB withdrawal.
  Interventions: Drug: Pentobarbital

INTERVENTIONS:
Drug: Lorazepam — Lorazepam
  Other Names: Ativan
  Arms: Lorazepam
Drug: Pentobarbital — Pentobarbital
  Other Names: Nembuta
  Arms: Pentobarbital

SUMMARY:
Gamma hydroxybutyrate (GHB) is a powerful central nervous system depressant. The number of individuals seeking treatment for GHB abuse has been steadily increasing in the United States. Currently, lorazepam and pentobarbital are two medications used to treat individuals who experience GHB-withdrawal symptoms. The purpose of this study is to describe the signs and symptoms of GHB withdrawal and to identify predictors of withdrawal severity. The study will also evaluate the safety and effectiveness of treatment with lorazepam versus pentobarbital for GHB detoxification.

DETAILED DESCRIPTION:
GHB and GHB precursors such as 1,4-butanediol and gamma-butylrolactone (GBL) have become popular drugs of abuse. In cases of severe withdrawal, delirium, confusion, hallucinations, and agitation can occur. There has been a sharp rise in the number of GHB related emergency room visits over the past few years, yet little is known about the effective treatment of GHB withdrawal and dependence. The purpose of this study is to describe the signs and symptoms of GHB withdrawal, identify predictors of withdrawal severity, and evaluate the safety and effectiveness of treatment for GHB detoxification. There will be compensation for screening assessments.

The study includes two phases. The open-label Phase 1 will aim to determine the safety of lorazepam for the treatment of mild GHB withdrawal. Participants who progress into moderate or severe withdrawal will enter the controlled Phase 2. In Phase 2, participants will be randomly assigned to receive either lorazepam or pentobarbital in order to determine which drug is more effective in treating GHB withdrawal.

The study will consist of 1 to 2 outpatient screening visits, followed by up to 15 days of inpatient detoxification treatment and assessment. After hospital discharge from inpatient treatment, measures of protracted GHB withdrawal and psychiatric symptoms will be obtained on an outpatient weekly basis for 8 weeks. Repeat measures of cognitive functioning will be obtained at baseline, termination of treatment, and at 30, 60, and 90-day follow-up intervals in order to assess long-term neurocognitive effects of GHB withdrawal and use.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for GHB dependence
* Self-reported as GHB dependent with current daily use of GHB
* Use of GHB for at least 20 consecutive days prior to enrollment
* Desire to stop GHB use
* Availability of a friend or family member to act as a collateral informant
* Speaks and understands English

Exclusion Criteria:

* Females who are pregnant, breastfeeding, or do not agree to use adequate forms of contraception
* History of seizures
* A baseline EEG of clinical concern that requires inpatient ICU detoxification
* Any anticonvulsant therapy during the 3 years prior to enrollment
* Pancreatic disease, such as insulin-dependent diabetes
* Liver disease that requires medication or medical treatment
* Gastrointestinal or kidney disease that might significantly impair absorption, metabolism, or excretion of study drug, or might require medication or medical treatment
* Asthma, hives, angioedema, or similar condition
* Acute intermittent porphyria or porphyria variegata
* Neurological or psychiatric disorders, including psychosis, bipolar disorder, or other disorders that require treatment or might make study compliance difficult (assessed by the Structured Clinical Interview for DSM-IV-TR)
* Positive tuberculosis (PPD) skin test with a clinical history and chest X-ray indicative of active tuberculosis (individuals with a positive PPD test and a negative chest X-ray, who are not symptomatic for tuberculosis and do not require antituberculosis therapy, will be eligible to participate)
* Clinically significant abnormal baseline EKG
* Requirement for any of the following medications currently or within the 4 weeks prior to enrollment: psychotropics (including sedatives/hypnotics, antidepressants, neuroleptics), prescription analgesics, anticonvulsants, antihypertensives, antiarrhythmics, or antiretroviral medications
* Nicotine dependent participants will be given nicotine patch therapy for the duration of the study; participants who refuse nicotine patch therapy will continue in the study as determined by the hospital smoking and standard of care regulations
* Meets DSM-IV criteria for dependence on any psychoactive substance other than GHB, caffeine, or nicotine
* Symptomatic HIV infection
* Alcohol breath test greater than .05 ppm at time of hospital admission

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2004-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Subjective withdrawl symptoms measures using CIWA scale | daily during medical administration

CONTACTS AND LOCATIONS:
Overall Officials: Karen Miotto, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

REFERENCES:
- See also: UCLA GHB Research Study — http://www.uclaisap.org/projects/miotto07A.html